CLINICAL TRIAL: NCT02438293
Title: 'The Impact of Rhinovirus Infections in Paediatric Cardiac Surgery'
Acronym: RISK
Status: Completed | Type: Observational
Sponsor: Leiden University (Other)
Responsible Party: Principal Investigator, JuttedeVries, M.D. PhD, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Other Study IDs: P14.303
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Rhinovirus; Congenital Heart Disease; Respiratory Infections; Post-operative Complications
Keywords: rhinovirus; cardiac surgery; paediatric; respiratory infection; children
MeSH Terms: conditions — Heart Defects, Congenital; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal swabs serum EDTA plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children undergoing cardiac surgery: paediatric patients with a congenital heart disease undergoing elective cardiac surgery
  Interventions: Other: rhinovirus diagnostics

INTERVENTIONS:
Other: rhinovirus diagnostics — rhinovirus PCR on a nasopharyngeal swab

SUMMARY:
This is a prospective single- center observational study in the Leiden University Medical Center in approximately 250 children (<12 years) undergoing elective cardiac surgery, for congenital heart disease. The parents/guardians of the children will be asked to fill out a questionnaire, to asses respiratory symptoms in the last weeks, before the operation of their child. In the operating theatre, a nasopharyngeal swab will collected. Clinical data will be collected daily during paediatric intensive care admission, and date of discharge from paediatric intensive care unit and from hospital are recorded. If children are still intubated at day 4 a second nasopharyngeal swab and residual blood will be collected. The samples will be tested for rhinovirus with a polymerase chain reaction. Main study parameter is the paediatric intensive care unit length of stay in per-operative rhinovirus -positive compared to rhinovirus-negative patients.

DETAILED DESCRIPTION:
Rationale:

Respiratory infections are considered to carry a potential risk of adverse events in children undergoing surgery.

Rhinovirus is a common cause of respiratory infections and congenital heart disease is a risk factor for severe rhinovirus infection. However, we do not know what the impact of clinical or subclinical rhinovirus infections is on postoperative course following congenital heart surgery in children.

Based on our clinical experience, one case-controlled study , and a case reported in the literature, we hypothesize that paediatric patients with per-operative rhinovirus positive Polymerase Chain Reaction (PCR) testing have a longer paediatric intensive care unit (PICU) admission , compared to children who test negative.

Objectives:

Primary: To identify whether PCR-proven rhinovirus is a risk factor for prolonged PICU admission in children undergoing cardiac surgery.

Secondary: to develop a preoperative algorithm to identify children with increased risk for prolonged PICU admission after cardiac surgery.

Study design:

This is a prospective single-center observational cohort study in the Leiden University Medical Center (LUMC).

Methods Parents of the selected patients will receive the information folder and a questionnaire by mail (asking for signs and symptoms of current and/or recent respiratory infections) when they receive the letter with the date of admission and operation.

On the day of admission (day -1) all (parents of) children admitted for cardiac surgery will be asked to participate in this study and fill out a written informed consent.

At day 0, the operation day, in the operating theatre a nasopharyngeal swab will be collected following anaesthetic induction and tested for rhinovirus. All clinicians will be blinded for the PCR results and will only be made known to the investigator from the virology department.

Clinical and laboratory data will be collected for all patients until discharge from the hospital. Of all the patients still on mechanical ventilation at day 4, an additional nasopharyngeal swab will be sampled and scavenge samples blood will be requested at the chemical laboratory if available. Rhinovirus PCR will be performed on nasopharyngeal swab and blood to determine shedding and viremia.

Residual blood (for infection parameters) will be collected at three time points: after induction of anaesthesia, directly after operation at PICU admission and at day four (4) when the patient is still on ventilator support.

ELIGIBILITY:
Inclusion Criteria:

* Children (<12 year) with a congenital heart disease undergoing elective cardiac surgery
* Written informed consent by parents or guardian

Exclusion Criteria:

* No informed consent from one of the parents (or the legal representative if applicable)
* Anaesthesiologist or cardiopulmonary surgeon postpones surgery based on routine hospital screening
* Emergency surgery
* Pre-operative admission to the neonatology department
* Children not admitted to the intensive care unit after cardiac surgery
* Children undergoing a second cardiac operation during the same intensive care stay
* Children with duct-dependent physiology who remain prostaglandin-dependent after the heart operation (they will be excluded because they will certainly have a prolonged PICU LOS regardless of a possible rhinovirus infection). For example: hypoplastic left heart syndrome following pulmonary artery banding who will remain on prostaglandins until the next staged operation

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (<12 year) with a congenital heart disease undergoing elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
post-operative PICU length of stay | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
  rhinovirus PCR positive compared to rhinovirus negative patients

SECONDARY OUTCOMES:
Duration of ventilatory support | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
mean airway pressure | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
FiO2 | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
peak inspiratory pressure (maximum values) | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
positive end expiratory pressure (maximum values) | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
Antibiotic free days (alive at PICU discharge) | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
Need of inotropes (inotrope score) | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
CRP | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
Leukocytes | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
Hospital length of stay | participants will be followed for the duration of PICU stay, an expected average of 3,8 days
Any secondary infection (bacterial, viral and parasitic infections) | participants will be followed for the duration of PICU stay, an expected average of 3,8 days

CONTACTS AND LOCATIONS:
Overall Officials: Anneloes L Klink, Msc, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Roeleveld PP, Van Rijn AL, de Wilde RBP, van Zwet EW, Wink J, Rozendaal L, Hogenbirk K, Hazekamp MG, Man WH, Sidorov I, Kraakman MEM, Claas ECJ, de Jonge E, Kroes ACM, de Vries JJC. Rhinovirus Detection in the Nasopharynx of Children Undergoing Cardiac Surgery Is Not Associated With Longer PICU Length of Stay: Results of the Impact of Rhinovirus Infection After Cardiac Surgery in Kids (RISK) Study. Pediatr Crit Care Med. 2021 Jan 1;22(1):e79-e90. doi: 10.1097/PCC.0000000000002522. PMID 33027243